CLINICAL TRIAL: NCT05735639
Title: THRomboprophylaxis in Individuals Undergoing Superficial endoVEnous Treatment (THRIVE) - a Multi-centre Assessor-blind Randomised-controlled Trial
Brief Title: THRomboprophylaxis in Individuals Undergoing Superficial endoVEnous Treatment (THRIVE)
Acronym: THRIVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22CX7510; ISRCTN18501431 (Other: ISRCTN)
Record Dates: First submitted 2023-01-19; First posted 2023-02-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Venous Thromboembolism; Varicose Veins
MeSH Terms: conditions — Venous Thromboembolism; Varicose Veins | interventions — Dalteparin; Tinzaparin; enoxaparin sodium; Rivaroxaban; apixaban; Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compression therapy alone (No Intervention)
- Compression therapy + single dose of low-molecular weight heparin at time of procedure (Experimental): A single prophylactic dose of low molecular weight heparin (LMWH) (e.g., dalteparin sodium, tinzaparin sodium, enoxaparin sodium) will be prescribed as per standard practice and administered in accordance with the relevant Summary of Product Characteristics (SmPC), manufacturer's recommendations and instructions for use.
  Interventions: Drug: Dalteparin Sodium; Drug: Tinzaparin Sodium; Drug: Enoxaparin Sodium
- Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC (Experimental): An extended duration of LMWH (e.g., dalteparin sodium, tinzaparin sodium, enoxaparin sodium) or an extended duration of a direct oral anticoagulant (DOAC) (e.g., rivaroxaban, apixaban, dabigatran etexilate) will be prescribed as per current local practice and administered in accordance with the relevant SmPC, manufacturer's recommendations and instructions for use. The duration of this must be at least 7 days, but can be in line with local practice i.e., 7, 10 or 14 days.
  Interventions: Drug: Dalteparin Sodium; Drug: Tinzaparin Sodium; Drug: Enoxaparin Sodium; Drug: Rivaroxaban; Drug: Apixaban; Drug: Dabigatran Etexilate

INTERVENTIONS:
Drug: Dalteparin Sodium — Low molecular weight heparin
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC; Compression therapy + single dose of low-molecular weight heparin at time of procedure
Drug: Tinzaparin Sodium — Low molecular weight heparin
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC; Compression therapy + single dose of low-molecular weight heparin at time of procedure
Drug: Enoxaparin Sodium — Low molecular weight heparin
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC; Compression therapy + single dose of low-molecular weight heparin at time of procedure
Drug: Rivaroxaban — Direct oral anticoagulant
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC
Drug: Apixaban — Direct oral anticoagulant
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC
Drug: Dabigatran Etexilate — Direct oral anticoagulant
  Arms: Compression therapy + single dose of LMWH at time of procedure + extended course of LMWH or DOAC

SUMMARY:
Endovenous interventions are keyhole operations for varicose veins that are carried out from within the vein itself. Varicose veins are enlarged veins close to the surface of the skin. They are connected to the bigger deeper veins in the leg (known as deep veins). Because of this, operations to close the varicose veins can increase the chance of a blood clot forming in the deep veins. Blood clots in the deep veins happen in around 1 in 50 people after endovenous operations. A clot in the leg can cause swelling, pain, and other long-term problems. If a clot in the leg breaks off and travels to the lungs, it can cause problems with the lung' ability to move oxygen from the air into the blood and may, in rare cases, be life threatening.

Varicose vein procedures may carry a slightly higher risk of blood clot formation, and we are currently unsure if current clot reducing medicines are beneficial in preventing blood clots in people having varicose vein procedures.

This study will investigate if it is worthwhile prescribing medicines to reduce blood clots after varicose vein procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Scheduled to undergo endovenous intervention of truncal varicose veins under local anaesthesia
* Treatment technologies including radiofrequency, laser, mechanochemical, foam sclerotherapy and cyanoacrylate glue

Exclusion Criteria:

* Clinical indication for therapeutic anticoagulation e.g., atrial fibrillation
* Previous personal or first-degree relative history of VTE
* Thrombophilia
* Female patients of childbearing potential who have a positive pregnancy test
* A history of allergy to heparins or direct oral anticoagulants
* A history of heparin-induced thrombocytopenia
* Inherited and acquired bleeding disorders
* Evidence of active bleeding
* Concomitant major health problems such as active cancer and chronic renal and/or liver impairment
* Known thrombocytopenia (platelets known to be less than 50 x 109

  /l)
* Surgery or major trauma in the previous 90 days
* Recent ischemic stroke in the previous 90 days
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6660 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging confirmed lower limb deep vein thrombosis (DVT) with or without symptoms, or pulmonary embolism (PE) with symptoms within 90 days of varicose vein treatment. | 90 days
  The rate of lower limb DVT with or without symptoms, or PE with symptoms within 90 days of varicose vein treatment.

SECONDARY OUTCOMES:
Lower limb DVT without symptoms | 21 - 28 days
  Duplex ultrasound scan
Lower limb DVT with symptoms | 90 days
  Self-reported VTE outcome questionnaire
PE with symptoms | 90 days
  VTE outcome questionnaire (self-reported) to determine the rate of PE
Comparisons of quality of life at 7- and 90-days post-procedure | 90-days
  Using EQ-5D
Cost-effectiveness of providing pharmacological thromboprophylaxis | 90 days
  Incremental Cost-Effectiveness Ratio (ICER)
Exploratory analyses to assess how well a VTE risk assessment tool predicts VTE outcome | 90 days
  Venous thromboembolism risk as determined by the Department of Health Risk Assessment tool
Exploratory analyses to assess how well a VTE risk assessment tool predicts VTE outcome | 90 days
  Venous thromboembolism risk as determined by the Caprini risk assessment model
Mortality rates in each group | 90 days
  Rate of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No